CLINICAL TRIAL: NCT07077785
Title: The Effects of Epidural Analgesia on Maternal-Infant Bonding and Birth-Related Trauma in Women Undergoing Vaginal Delivery With Epidural Analgesia
Brief Title: The Effects of Epidural Analgesia on Maternal-Infant Bonding and Birth-Related Trauma
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Adiyaman University Research Hospital (Other)
Responsible Party: Principal Investigator, Nezir Yılmaz, Assoc. Prof., Adiyaman University Research Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: ADYU-ANS-NY-011
Record Dates: First submitted 2025-07-12; First posted 2025-07-22 (Actual); Last update posted 2025-07-22 (Actual); Status verified 2025-07

CONDITIONS: Epidural Anesthesia in Labor and Delivery
Keywords: epidural analgesia; maternal-infant bonding; Psychological Birth Trauma
MeSH Terms: interventions — Analgesia, Epidural

STUDY DESIGN:
Intervention Model Description: This is a prospective, randomized, single-center, parallel-group clinical study designed to evaluate the psychological impact of epidural analgesia on childbirth-related outcomes. The study will compare two groups of women undergoing vaginal delivery: those receiving epidural analgesia and those not receiving it. Outcomes such as perceived pain (VAS), maternal satisfaction, psychological stress related to childbirth, and early maternal-infant bonding will be assessed through validated scales administered during hospitalization and at 1-month postpartum.
Who Masked: Investigator, Outcomes Assessor
Masking Description: Outcome assessors and data analysts will be blinded to group allocation. Although study participants and clinical staff involved in labor management are aware of the intervention status, the researchers who administered epidural analgesia will not participate in data collection or outcome evaluation. Therefore, the evaluation of questionnaire responses and study outcomes will be conducted independently, without knowledge of the participants' group assignment, ensuring assessor-level blinding.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Epidural group- group E (Experimental): Participants in this group will receive epidural analgesia during vaginal delivery
  Interventions: Procedure: Epidural Analgesia
- Control group- group C (No Intervention): Participants in this group will undergo vaginal delivery without receiving any form of neuraxial analgesia.

INTERVENTIONS:
Procedure: Epidural Analgesia — After informed consent and exclusion of contraindications, an epidural catheter will be placed at the L3-L4 interspace in the sitting position using a Tuohy needle. A test dose of 2 mL lidocaine will be administered to confirm correct catheter placement under continuous monitoring of vital signs. Once cervical dilatation reaches 5 cm, 5 mL of 0.2% bupivacaine combined with 25 mcg fentanyl will be administered via the epidural catheter. Additional boluses will be given as needed based on pain assessment. The catheter will be removed 24 hours postpartum.
  Arms: Epidural group- group E

SUMMARY:
This prospective, single-center study aims to evaluate the effects of epidural analgesia on maternal-infant bonding and perceived birth-related trauma in women undergoing vaginal delivery. Participants will be divided into two groups: those who receive epidural analgesia and those who deliver without it. Standardized questionnaires will be used to assess pain perception, maternal satisfaction, and the quality of early bonding between mother and infant. The study is designed in accordance with the Declaration of Helsinki and Good Clinical Practice guidelines, with approval from the local ethics committee.

DETAILED DESCRIPTION:
This study is a prospective, non-interventional, single-center clinical trial that will be conducted at Adıyaman University Training and Research Hospital, Department of Obstetrics and Gynecology. The aim is to investigate the impact of epidural analgesia on maternal-infant bonding and birth-related psychological trauma among women undergoing spontaneous vaginal delivery.

Eligible participants will include pregnant women aged between 18 and 40 years with ASA physical status I or II, who are planning vaginal delivery. Women with contraindications to epidural analgesia, morbid obesity, previous local anesthetic toxicity, or indications for cesarean section will be excluded.

Based on a priori power analysis, 40 participants will be recruited into each group to account for potential dropout, totaling 80 participants. Group E will consist of women who receive epidural analgesia during labor, while Group C will include those who undergo vaginal delivery without any epidural intervention.

Epidural analgesia will be administered via catheter placement at the L3-L4 vertebral level. Following a test dose with lidocaine, patients will receive a combination of 0.2% bupivacaine and 25 mcg fentanyl once cervical dilatation reaches 5 cm. Additional boluses may be administered as required based on pain levels.

Participants will be assessed for pain intensity using the Visual Analog Scale (VAS) during and after delivery. Postpartum satisfaction and early breastfeeding status will be recorded prior to discharge. At one month postpartum, all participants will complete validated questionnaires, including a birth-related trauma scale and the Maternal Attachment Inventory, to assess psychological outcomes and maternal-infant bonding.

The results of this study are expected to contribute to a better understanding of the psychological and emotional consequences of epidural analgesia in vaginal deliveries and help optimize maternal care practices.

ELIGIBILITY:
Inclusion Criteria:

Female participants aged between 18 and 40 years

ASA physical status classification I or II

Pregnant women undergoing spontaneous vaginal delivery at the study hospital

Willingness to provide informed consent and participate in study procedures

Exclusion Criteria:

Age below 18

ASA physical status classification III or IV

Morbid obesity (BMI ≥ 40 kg/m²)

Indication for cesarean section

History of local anesthetic toxicity or allergy

Contraindications to epidural analgesia (e.g., coagulopathy, infection at insertion site)

Any significant maternal or fetal complication that contraindicates study participation

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Only female participants who are pregnant and undergoing vaginal delivery will be eligible for inclusion in this study.
Enrollment: 80 (Estimated)
Dates: Start 2025-07-25 (Estimated); Primary Completion 2025-08-30 (Estimated); Study Completion 2025-09-15 (Estimated)

PRIMARY OUTCOMES:
Effect of Epidural Analgesia on Maternal-Infant Bonding Quality and Birth-Related Psychological Stress | 1 month postpartum
  Assessment of maternal-infant bonding quality using the Maternal Attachment Inventory (MAI) and evaluation of birth-related psychological stress using a validated childbirth trauma scale. Outcomes will be measured via structured questionnaires administered at 1 month postpartum to evaluate the psychological impact of epidural analgesia during vaginal delivery.

SECONDARY OUTCOMES:
Pain Intensity During Labor Assessed by Visual Analog Scale (VAS) | From labor onset until discharge (approximately 0 to 48 hours postpartum)
  Evaluation of maternal pain intensity during labor using the Visual Analog Scale (VAS). Pain scores will be recorded at predefined intervals, including active labor and immediately postpartum.

OTHER OUTCOMES:
Maternal Satisfaction with the Birth Experience | Within 48 hours postpartum (prior to discharge)
  Assessment of maternal satisfaction regarding the childbirth process using a validated satisfaction questionnaire administered prior to hospital discharge.

CONTACTS AND LOCATIONS:
Locations (1):
- Adıyaman University Training and Research Hospital, Adıyaman, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided